CLINICAL TRIAL: NCT02588339
Title: A Phase II Trial Evaluating the Use of a Histone Deacetylase Inhibitor Panobinostat for Graft Versus Host Disease (GVHD) Prevention
Brief Title: Panobinostat (LBH589): Acute Graft Versus Host Disease (aGVHD) Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-18374; CLBH589US100T (Other: Novartis)
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Graft Versus Host Disease; GVHD
Keywords: Hematologic disorder; allogeneic hematopoietic cell transplantation
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Diseases | interventions — Panobinostat; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat (PANO) Therapy (Experimental): Participants will be treated with standard of care chemotherapy agents prior to their allogeneic hematopoietic cell transplant. For Graft Versus Host Disease (GVHD) prevention, participants will receive PANO, Sirolimus and Tacrolimus.
  Interventions: Drug: Panobinostat; Drug: Sirolimus; Drug: Tacrolimus

INTERVENTIONS:
Drug: Panobinostat — Panobinostat (PANO) will begin 5 days (Day -5) before transplant day (Day 0). All participants will take PANO by mouth once a day, three times a week (48 hours apart), every week for 26 weeks (approximately 6 months). PANO will be provided by Novartis as 5-mg pink gelatin capsules.
  Other Names: PANO; Farydak; LBH-589
Drug: Sirolimus — Sirolimus will be given the day before transplant and continued daily for at least one year. SIR will be administered starting on day -1 and thereafter. Dosing will be adjusted to maintain therapeutic targets per Moffitt institutional standards.
  Other Names: SIR; Rapamune
Drug: Tacrolimus — Tacrolimus as an infusion or as a pill will begin 3 days before transplant (day -3) and following Moffitt institutional guidelines for dosing. Tacrolimus will be given for at least 50 days and participants will remain on Tacrolimus for as long as it is necessary per standard of care.
  Other Names: TAC; Prograf

SUMMARY:
This study will test PANO in combination with tacrolimus/sirolimus (TAC/SIR) for acute GVHD prevention. The purpose of this study is to determine if Panobinostat (PANO) when used in combination with sirolimus and tacrolimus will help reduce the incidence of Graft-vs-host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older at time of enrollment
* Signed informed consent
* Hematologic disorder requiring allogeneic hematopoietic cell transplantation
* Left ventricular ejection fraction (LVEF) ≥ 45% by multiple uptake gated acquisition (MUGA) scan or echocardiogram
* Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and diffusing lung capacity oxygenation (DLCO) adjusted ≥ 50% of predicted values on pulmonary function tests
* Transaminases (AST, ALT) < 3 times upper limit of normal (ULN) values
* Creatinine clearance calculated ≥ 50 mL/min
* Karnofsky Performance Status Score ≥ 60%.
* Human leukocyte antigen (HLA) matched 8/8 (A, B, C, DRB1) related or unrelated donor

Exclusion Criteria:

* Active infection not controlled with appropriate antimicrobial therapy
* HIV, hepatitis B (HBcAb positive but HBsAg negative with undetectable viral load are eligible), or hepatitis C infection
* Sorror's co-morbidity factors with total score > 4. Important modification to co-morbidity index calculation: DLCO adjusted will not be included in assessment of pulmonary risk, except those patients with DLCO adjusted < 50% who are excluded from the trial.
* Anti-thymocyte globulin (ATG) as part of the conditioning regimen
* Cyclophosphamide as part of the conditioning regimen or for GVHD prophylaxis
* Pregnancy
* Histone deacetylase (HDAC), DAC, HSP90 inhibitors or valproic acid for the treatment of cancer within 30 days
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first PANO treatment
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following: Any history of ventricular fibrillation or torsade de pointes; Bradycardia defined as heart rate (HR)< 45 bpm (Patients with pacemakers are eligible if HR ≥ 45 bpm); Screening electrocardiogram (ECG) with a QTcF > 480 msec; Right bundle branch block + left anterior hemiblock (bifascicular block); Patients with myocardial infarction or unstable angina ≤ 12 months prior to starting study drug; Other clinically significant heart disease (e.g., New York Heart Association (NYHA) class III or IV , uncontrolled hypertension) as per discretion of principal investigator and/or treating physician; Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug with the exception of drugs listed on Appendix B of study documents that are required for hematopoietic cell transplantation (HCT) patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lia Perez, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Lakshmanan AP, Deola S, Terranegra A. The Promise of Precision Nutrition for Modulation of the Gut Microbiota as a Novel Therapeutic Approach to Acute Graft-versus-host Disease. Transplantation. 2023 Dec 1;107(12):2497-2509. doi: 10.1097/TP.0000000000004629. Epub 2023 May 16. PMID 37189240
- [Derived] Perez L, Fernandez H, Kharfan-Dabaja M, Khimani F, Betts B, Mishra A, Ayala E, Locke FL, Ochoa-Bayona L, Nieder M, Pidala J, Achille A, Powers J, Sahakian E, Thapa R, Wang X, Anasetti C. A phase 2 trial of the histone deacetylase inhibitor panobinostat for graft-versus-host disease prevention. Blood Adv. 2021 Jul 13;5(13):2740-2750. doi: 10.1182/bloodadvances.2021004225. PMID 34242388
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between March 2016 and August 2018
Groups:
- Panobinostat (PANO) Therapy: Participants treated with standard of care chemotherapy agents prior to their allogeneic hematopoietic cell transplant. For Graft Versus Host Disease (GVHD) prevention, participants received PANO, Sirolimus and Tacrolimus. GVHD graded using NIH criteria, scores of 0-3 per area of involvement (e.g; skin, liver and gut) 0 being no symptoms and 3 being symptomatic, over 50% of waking hours in bed, ECOG 3-4.
Period: Overall Study
Arm/Group | Panobinostat (PANO) Therapy
Started | 42
Completed | 39
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — GVHD Progression prior to treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Panobinostat (PANO) Therapy
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 58 [19 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 36
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Stratified by Acute Graft Versus Host Disease GVHD Stage
Description: Cumulative incidence of acute GVHD grades II-IV by day 100. Investigators will consider ≥43% incidence of grade II-IV aGVHD not acceptable. Investigators will use 23% incidence rate of GVHD as target. GVHD severity stage and grading and distribution will be measured weekly from day of transplant to day 90 +/- 14 using standard scoring system. Stage of GVHD will be given for each site of involvement (e.g. skin, liver, and gut), as well as a composite score for overall acute GVHD grade. Pathologic confirmation of aGVHD will be dictated by usual clinical practice, and not mandated by this protocol.
Time Frame: 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat (PANO) Therapy
Number analyzed (Participants) | 7
Participants
  Grade II GVHD | 6
  Grade III GVHD | 1

2. Secondary Outcome: Number of Participants Stratified by Chronic Graft Versus Host Disease (GVHD) Stage
Description: GVHD with onset after 100 days post-HCT with presence of at least one diagnostic manifestation of chronic c-GVHD or distinct manifestation confirmed by biopsy or other relevant tests (e.g., PFT). Classified as: 1- Classic chronic GVHD - meets criteria for chronic GVHD and has no features consistent with aGVHD or 2-Overlap syndrome - features of acute and chronic GVHD exist together. C-GVHD will be measured prospectively in all participants on days 90+/-14 , 120 +/- 14, 150 +/- 14, 180+/- 14, 270+/- 30, and 365 +/- 30 as per standardized scoring system.
Time Frame: 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat (PANO) Therapy
Number analyzed (Participants) | 12
Participants
  Mild GVHD | 10
  Moderate GVHD | 2

3. Secondary Outcome: Time to Stable Engraftment
Description: Stable engraftment for white blood count (WBC) is defined as a sustained absolute neutrophil count > 500 over 3 days without cytokine support. Stable platelet engraftments is defined as count of > 20,000 over 7 days without transfusion support. Time to engraftment is defined as time from day 0 to day of sustained engraftment per above criteria for both platelets and WBC.
Time Frame: 100 days post transplant
Population: Participants with stable engraftment were analyzed
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Panobinostat (PANO) Therapy
Number analyzed (Participants) | 38
days
  ANC engraftment | 15 [12 to 21]
  Platelet engraftment | 16 [9 to 31]

4. Secondary Outcome: Number of Participants With Primary Disease Relapse
Description: Incidence of primary disease relapse and non-relapse related death will be reported per standard definitions. These will be treated as competing risk events.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat (PANO) Therapy
Number analyzed (Participants) | 39
Participants | 7

5. Secondary Outcome: Number of Participants With Non-relapse Mortality
Description: Incidence of primary disease relapse and non-relapse related death will be reported per standard definitions. These will be treated as competing risk events. Non-relapse death is defined as death in continuous remission from primary disease requiring transplantation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat (PANO) Therapy
Number analyzed (Participants) | 39
Participants | 1

6. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Overall survival: Time from transplant date to death from any cause. Time-to-event data such as overall survival is measured from the date of transplantation. OS will be analyzed using the Kaplan-Meier method.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Panobinostat (PANO) Therapy
Number analyzed (Participants) | 39
percentage of participants | 87

7. Secondary Outcome: Percentage of Participants With Relapse-free Survival (RFS)
Description: Relapse-free survival: Time from transplant date to death or primary disease relapse. Time-to-event data such as relapse-free survival is measured from the date of transplantation. RFS will be analyzed using the Kaplan-Meier method.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Panobinostat (PANO) Therapy
Number analyzed (Participants) | 39
percentage of participants | 77

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Arm/Group | Panobinostat (PANO) Therapy
All-Cause Mortality (participants affected / at risk) | 2/39
Serious Adverse Events (participants affected / at risk) | 12/39
Other Adverse Events (participants affected / at risk) | 32/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat (PANO) Therapy (N=39)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders -Other (Skin and subcutaneous tissue disorders) | 1 (1) — skin infection
Confusion (Psychiatric disorders) | 2 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Immune system disorders -Other (Immune system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (2)
Aspartate aminotransferase increased -Transiminitis (Investigations) | 1 (2)
Hepatobiliary disorders - other (Hepatobiliary disorders) | 2 (3)
Appendicitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat (PANO) Therapy (N=39)
Lung Infection (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Encephalitis infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 10 (12)
Non-cardiac chest pain (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 7 (9)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Myelitis (Nervous system disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Floaters (Eye disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Akathisia (Nervous system disorders) | 2 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Immune system disorders -Other (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02588339/Prot_SAP_000.pdf